CLINICAL TRIAL: NCT05604755
Title: Effect of Prophylactic HQP1351 Maintenance Post-transplants on Ph+ Luekemia Undergoing Allo-HSCT With MRD Positive Pre-transplants
Brief Title: Prophylactic HQP1351 Therapy Post-transplants on Leukemia After Allo-HSCT
Acronym: Case-Only
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Drugs was too expensive eligible for inclusion
Sponsor: xuna (Other)
Collaborators: Nanfang Hospital, Southern Medical University (Other); Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Second Provincial General Hospital (Other)
Responsible Party: Sponsor-Investigator, xuna, professor, Nanfang Hospital, Southern Medical University
Organization: Nanfang Hospital, Southern Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PH20221030
Record Dates: First submitted 2022-10-30; First posted 2022-11-03 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Prophylactic HQP1351 Therapy; Third Generation TKI
Keywords: CML; ph+ ALL; HQP1351; Prophylactic therapy
MeSH Terms: interventions — olverembatinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HQP1351 prophylactic therapy (Experimental): HQP1351 prophylactic therapy after allo-hct on days 30 to 60
  Interventions: Drug: HQP1351( Olverembatinib dimesylate)

INTERVENTIONS:
Drug: HQP1351( Olverembatinib dimesylate) — HQP1351 was initiated at a dose of 40mg every two days

SUMMARY:
Allogeneic hematopoietic stem cell transplantation (allo-HSCT) improves the long-term outcomes for Philadelphia chromosome-positive acute lymphoblastic leukemia (Ph+ ALL) and BC-CML. Relapse remains a major cause of treatment failure even after allo-HSCT. The prevention of relapse is essential for improving the outcome of Ph+ ALL. Pre-emptive tyrosine kinase inhibitor (TKIs) administration based on minimal residual disease (MRD) and BCR-ABL mutation after allo-HSCT might reduce the incidence of relapses and improve survival for patients with Ph+ luekemia. In this study, we will evaluate the safety and efficacy of newly third TKI-HQP1351 therapy post-transplants on Ph+ leukemia after allo-HSCT with MRD positive pre-transplants.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age of 18-65 years
2. Ph+ luekemia(includ Ph+ALL and CML) undergoing allo-HSCT with MRD positive pre-transplants
3. Survival > 30 days post-transplants
4. Laboratory parameters as defined below:

   Serum creatinine less than or equal to 2.0 x ULN AST and ALT less than or equal to 3 x ULN (less than or equal to 5 x ULN if unequivocal liver GvHD),Total bilirubin less than or equal to 3 x ULN
5. Ability to understand and willingness to sign a written informed consent form

Exclusion Criteria:

1. Ph+ ALL undergoing allo-HSCT with MRD negative pre-transplants
2. Survival <30 days post-transplants
3. MRD positive on day +30 post-transplants
4. Any abnormality in a vital sign (e.g., heart rate, respiratory rate, or blood pressure)
5. Patients with any conditions not suitable for the trial (investigators' decision)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival（DFS） | 2 years
  The time from the date of transplantation to leukemia relapse

SECONDARY OUTCOMES:
Overall survival(OS) | 2 years
  the time from the date of transplantation to relapse or death or the last day of follow-up the time from the date of transplantation to relapse or death or the last day of follow-up the time from the date of transplantation to relapse or death or the last day of follow-up the time from the date of transplantation to relapse or death or the last day of follow-up the time from the date of transplantation to relapse or death or the last day of follow-up the time from the date of transplantation to relapse or death or the last day of follow-up The time from the date of transplantation to death or the last day of follow-up
Relapse rate | 2 years
  the cumulative relapse rate of leukemia
Adverse effects of TKI therapy | 2 years
  Number of participants with treatment-related adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Hematology, Nanfang Hospital, Southern Medical University,, Guanzhou, China

IPD SHARING:
Plan to Share IPD: No